CLINICAL TRIAL: NCT06574191
Title: The Effects of Patient and Visit Characteristics on Health Outcomes in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michelle Dossett, Associate Professor in Residence, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2054088; R01AG078283 (NIH)
Record Dates: First submitted 2024-05-15; First posted 2024-08-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diclofenac (Experimental): All study participants receiving topical diclofenac gel 1%. Participants will be instructed to apply 4 grams of the gel to the index knee at least once per day, and up to 4 times per day, for 8 weeks.
  Interventions: Drug: Topical Diclofenac gel 1%

INTERVENTIONS:
Drug: Topical Diclofenac gel 1% — Topical NSAID

SUMMARY:
The goal of this clinical trial is to understand the patient and clinic visit characteristics that affect health outcomes for individuals with knee osteoarthritis (OA) pain using topical diclofenac gel. The main questions it aims to answer are:

* What baseline patient characteristics predict response to topical diclofenac?
* Does patient physiology during the study visit predict response to topical diclofenac?
* Do study visit characteristics predict response to topical diclofenac?

Participants will:

* attend 2 study visits to complete study questionnaires and have blood drawn
* apply topical diclofenac to their knee for 8 weeks
* complete biweekly questions about knee pain and diclofenac use between study visits

DETAILED DESCRIPTION:
220 older adults with symptomatic knee OA will attend a single research clinic visit (one of four different types of study visits) with a study clinician. The investigators will video record the visits and measure participant heart rate and skin conductance during the visit. Participants will complete baseline questionnaires immediately prior to the study visit. All participants will receive diclofenac gel (a topical over-the-counter non-steroidal anti-inflammatory drug [NSAID]), a guideline recommended treatment for knee OA-related pain at the end of the first study visit. Participants will identify an "index" knee (worst pain, right or left) that they will treat and follow during the study. Between study visit 1 and the 8-week follow-up visit, participants will receive an every other week text message asking them to report on pain and diclofenac use to better understand changes in pain over time. Final questionnaires will be completed at the second study visit at week 8.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 50 years of age or older
* Radiographically confirmed knee OA of K/L grade 2 or higher within the past 2 years
* Knee pain at least 15 days/month.
* Average worst daily pain 3/10 or higher over a two-week period.

Exclusion Criteria:

* Medical contraindication to taking NSAIDs such as: history of coronary artery bypass graft, myocardial infarction, coronary artery stent placement, or stroke within the past 6 months; systolic heart failure with ejection fraction <45%; chronic kidney disease stage ≥4; severe gastrointestinal bleed or stomach ulcer within the past 6 months; current pregnancy; cirrhosis; currently taking blood thinners (aspirin 81 mg daily is okay); allergy to NSAIDs or aspirin; or any other medical contraindication to using topical NSAIDs.
* Inflammatory arthritis
* Partial or total knee replacement of the index knee
* Recent therapeutic injection of the index knee (less than 12 weeks)
* Planned knee/lower limb surgery during the two-month study period
* Active cancer treatment not in remission or life expectancy less than 6 months
* Inability to provide informed consent (e.g. dementia)
* Current use of topical or oral NSAIDs more than 3 days per week.
* Inability to receive text messages or emails to complete questionnaires between study visits.
* Unable to follow the study protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2028-01-27 (Estimated); Study Completion 2028-01-27 (Estimated)

PRIMARY OUTCOMES:
Knee Pain | 8 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) pain score from the index knee at 8 weeks. Score range 0-20. Higher scores signify worse pain.
Knee Function | 8 weeks
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) physical function score from the index knee at 8 weeks. Score range 0-68. Higher scores signify worse function.

SECONDARY OUTCOMES:
Global Impressions | 30 minutes
  Baseline-adjusted end of visit global impression ratings from study visit video recordings. Each global impression is measured on a 1-9 scale. Global impressions include engagement (clinician and patient), friendliness (clinician and patient), relaxed (clinician and patient), empathic (clinician), reciprocity (dyad), business-like (clinician), dominant (clinician), rushed/hurried (clinician), bored/uninterested (clinician), confident (patient), and pleased (patient). We will construct a Global Impression Summative Scale Score if a preliminary round of psychometric evaluation determines that a combination of the individual construct scores can be constructed that has adequate internal consistency and unidimensionality.
Non-verbal Behaviors | 30 minutes
  Baseline-adjusted end of visit non-verbal behaviors from study visit video recordings. Each non-verbal behavior is measured as counts (number of times) or total length of time within a discrete period of time (i.e., 2 minutes) from the video. Nonverbal behaviors that will be counted or timed for both parties include: gaze duration and number, smile duration and number, number of nods, self-touch, and gestures. We will also assess the number of clinician backchannel responses while patients spoke, the number of instances of shared laughter between the dyads, and the length of time that both the patient and clinician spoke. We will construct a Non-verbal Behavior Summative Score if a preliminary round of psychometric evaluation determines that a combination of the individual construct scores can be constructed that has adequate internal consistency and unidimensionality.
Skin conductance index measure | 30 minutes
  Concordance in skin conductance response (measured in micro Siemens) from electrodes attached to the patient's and clinician's fingers over the course of the study visit will be calculated using an established approach (Marci CD, 2007; PMID 17299296) to create a single index value for the visit. The natural logarithm of this value will be taken to reduce skew. A value greater than 0 means more than 50% concordance in the data, a value less than zero means less than 50% concordance in the data.
Change in patient skin conductance response | 30 minutes
  Change in patient skin conductance response from beginning to end of the initial study visit in micro-Siemens as measured by skin electrodes. Change score will be calculated as mean skin conductance response for the first 2 minutes of the study visit minus the mean value for the last 2 minutes of the study visit.
Heart rate variability index measure | 30 minutes
  Concordance in heart rate variability, measured from electrodes attached to the patient and clinician, over the course of the study visit, will be calculated using established approaches (see references below). Concordance is quantified by the degree to which heart rate variability of the patient and clinician are "in-phase" or "anti-phase" linked (i.e., coordinated changes in the same or opposite direction) along the study visits.
  https://pubmed.ncbi.nlm.nih.gov/29683720/ https://pubmed.ncbi.nlm.nih.gov/21910541/ https://pubmed.ncbi.nlm.nih.gov/24708502/ https://pubmed.ncbi.nlm.nih.gov/35315937/
Change in patient RMSSD (root mean square of successive differences) | 30 minutes
  The RMSSD component (proxy for high frequency heart rate variability) will be measured in the patient over the course of the study visit. Change score will be calculated as mean RMSSD value for the first 5 minutes of the study visit minus the mean value for the last 5 minutes of the study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Dossett, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified questionnaire and COMT genotype data will be available upon reasonable written request after publication and upon completing a data transfer agreement. Raw video and physiologic data will not be shared due to participant confidentiality/privacy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following publication of those data.
Access Criteria: Completion of a data transfer agreement.